CLINICAL TRIAL: NCT01490775
Title: Pilot Study to Assess Telemonitoring of Gleevec (Imatinib Mesylate) or Tasigna (Nilotinib)Therapy
Brief Title: Pilot Study to Assess Telemonitoring of Gleevec (Imatinib Mesylate) or Tasigna (Niltinib) Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to lack of funding
Sponsor: Rex Cancer Center, Raleigh, NC (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CAMN107AUS12T
Record Dates: First submitted 2011-10-14; First posted 2011-12-13 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2017-04

CONDITIONS: Chronic Phase CML
Keywords: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eMedonline access (Experimental): patients will be followed for 3 months with access to eMedonline
  Interventions: Behavioral: eMedonline access
- no access to eMedonline (Active Comparator): patients will be followed for 3 months with no access to eMedonline
  Interventions: Behavioral: no access to eMedonline

INTERVENTIONS:
Behavioral: no access to eMedonline — patients will be followed for 3 months but will not use eMedonline
  Other Names: Telemonitoring system; e-diary; electronic diary
  Arms: no access to eMedonline
Behavioral: eMedonline access — patients will be given access to eMedonline use for 3 months
  Other Names: Telemonitoring system; e-diary; electronic diary
  Arms: eMedonline access

SUMMARY:
This study is being conducted in a population of patients with chronic phase Chronic Myeloid Leukemia (CML) to learn more about how patients follow prescribed regimens for taking oral cancer drugs.

DETAILED DESCRIPTION:
This is a randomized, controlled pilot study to introduce eMedonline telemonitoring technology to CML patients taking Gleevec or Tasigna. eMedonline will be used to automatically collect time-dose specific medication data for individual patients, including dosing times, missed doses, adverse events and e-diary data. All data will be available to research staff for remote review via Web interface. Adverse events and non-adherence will prompt interventions including supportive care counseling.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older.
* Pathologically documented diagnosis of Chronic Phase CML (Ph+) in whom treating physician has determined that treatment with imatinib or nilotinib is appropriate
* Patients currently receiving Gleevec (imatinib) 300-600 mg daily or Tasigna (nilotinib) 300-400 mg twice daily
* Known performance status 0,1 or 2 (ECOG)
* Known adequate end organ function, defined as:

Total bilirubin < 1.5 xULN SGOT and SGPT <2.5 x ULN ANC > 1.5 Platlets > 100,000

* Patient is willing and able to use a cell phone
* Written, voluntary informed consent

Exclusion Criteria:

* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-04; Primary Completion 2015-02-12 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
eMedonline will be used to measure non-compliance in taking oral drug regimens. | at 6 months, non-compliance will be measured in each arm of study
  Patients are stratified to one of two groups: Group 1 is pateints on Gleevec or Tasigna who have been on drug less than 6 months; Group 2 is patients on Gleevec or Tasigna who have been on drug for equal to or more than 6 months.
  Group 1 is then divided into 2 groups: one using eMedonline for 3 months and the other not using eMedonline for 3 months. A crossover survey and pill counts will be done at the 3 month timepoint and then the groups will switch their access status to eMedonline.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wehbie, MD, Principal Investigator — Rex Cancer Center - Wakefield
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Rex Cancer Center - Wakefield, Raleigh, North Carolina